CLINICAL TRIAL: NCT05356767
Title: the Director of Vascular Surgery of Hospital of Chengdu University of Traditional Chinese Medicine
Brief Title: The Study of Percutaneous Mechanical Thrombectomy Treating Acute Deep Vein Thrombosis of Lower Extremities
Status: Recruiting | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, the director of the vascular surgery of Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Other Study IDs: ChengduUTCMvs3
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Pharmacomechanical Thrombolysis; Deep Vein Thrombosis
Keywords: Pharmacomechanical thrombolysis; Deep vein thrombosis; post-thromboticsyndrome
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post-thromboticsyndrome: suffering from PTS (Villalta score) at 2 years after operation.
  Interventions: Procedure: Pharmacomechanical thrombolysis
- n-post-thromboticsyndrome: none of PTS (Villalta score) at 2 years after operation.
  Interventions: Procedure: Pharmacomechanical thrombolysis

INTERVENTIONS:
Procedure: Pharmacomechanical thrombolysis — Pharmacomechanical thrombolysis

SUMMARY:
This study is a prospective, multicenter, real world, observational study intended to understand tmechanical thrombectomy in the treatment of acute deep venous thrombosis of lower extremities, It is estimated that 600 patients with DVT were enrolled in the group at 24 centers nationwide from May 2022 to May2024. we can obtain data on the incidence of sequelae of deep venous thrombosis after PMT, and analyze the factors that may affect the efficacy of PMT.

DETAILED DESCRIPTION:
Through inclusion and exclusion criteria, 600 patients were collected. This experiment was an observational study case series, and no control group was established. The patency of the lower extremity veins was assessed by lower extremity venous ultrasound or lower extremity venography. According to the postoperative symptoms and signs of the patients, the Villata score, (VEINS QoL)/Sym questionnaire and VCSS score were used to understand the PTS situation.Postoperative clinical follow-up was performed at 6 months, 12 months, 18 months, and 24 months. The main endpoints were the patency rate of lower extremity deep veins at 6 months after operation and the incidence of PTS (Villalta score) at 2 years after operation.

ELIGIBILITY:
Inclusion Criteria:

1. The symptoms of deep venous thrombosis of lower extremities occurred within 14 days (including 14 days)；
2. Lower extremity deep venous thrombosis involving iliac vein or / and femoral vein ;
3. Obtain the informed consent of all patients.

Exclusion Criteria:

1. Patients with a previous history of ipsilateral proximal lower limb deep venous thrombosis ;
2. patients who are prohibited from thrombolytic therapy;
3. inferior vena cava compression syndrome；
4. Allergic to heparin, low molecular weight heparin or contrast medium;
5. Patients who have participated in clinical trials of other drugs or medical devices that interfere with this clinical trial in the past 3 months;
6. Patients who do not want to participate in this trial;
7. Patients with poor compliance, or those who the researchers think are not suitable for selection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Deep vein thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Lower extremity deep vein patency rate 6 months after operation | 6 months
  The patency of the lower extremity veins was assessed by lower extremity venous ultrasound or lower extremity venography.
Incidence of sequelae of deep venous thrombosis after PMT | 24 months
  According to the postoperative symptoms and signs of the patients, the Villata score, (VEINS QoL)/Sym questionnaire and VCSS score were used to understand the PTS situation.

SECONDARY OUTCOMES:
Total duration of interventional treatment | 1 day
  Including the entire operation time of interventional surgery
Total urokinase dosage | 1 day
  interventional surgery urokinase dosage
Lower extremity deep venous patency rate of patients before discharge | 1 week
  The patency rate of lower extremity deep veins in patients 1 week after operation
Postoperative quality of life score (QOL) | 6 months,12 months,18 months and 24 months
  Postoperative quality of life scoring using the QOL scale
reoperation rate | 6 months,12 months,18 months and 24 months
  Reoperation due to thrombosis, pts
Incidence of bleeding complications | 1day，7day，3 months
  Symptoms of perioperative hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ye, doctor, Principal Investigator — Study Principal Investigator RenJi Hospital; Ziheng Wu, doctor, Principal Investigator — Study Principal Investigator Zhejiang University; Lianrui Guo, doctor, Principal Investigator — Study Principal Investigator Xuanwu Hospital, Beijing; Xin Fang, doctor, Principal Investigator — Study Principal Investigator Hangzhou first people's Hospital of Medical College of Zhejiang University; Hongfei Sang, doctor, Principal Investigator — Study Principal Investigator Second Affiliated Hospital of Suzhou University; Qiang Li, doctor, Principal Investigator — Study Principal Investigator Qingdao Haici Hospital affiliated to Qingdao University; Zibo Feng, doctor, Principal Investigator — Study Principal Investigator Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology; Zhenyu Shi, doctor, Principal Investigator — Shanghai Zhongshan Hospital; Weihao Shi, doctor, Principal Investigator — Huashan Hospital; Wensheng Lou, doctor, Principal Investigator — The First Affiliated Hospital With Affiliated Nanjing Medical University; Hui Zhao, doctor, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Chunshuihe, Chengdu, Sichuan, China